CLINICAL TRIAL: NCT06109103
Title: Investigation of the Effects of Telerehabilitation-based Motor Imagery Training on Motor Imagery Skills, Motor Function and Physical Performance in Children With Duchenne Muscular Dystrophy
Brief Title: Telerehabilitation-based Motor Imagery Training in Children With Duchenne Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Bora, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22114
Record Dates: First submitted 2023-06-19; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Telerehabilitation-based physiotherapy program + telerehabilitation-based motor imagery training Telerehabilitation-based physiotherapy program; Eight (8) weeks, three (3) sessions per week, 40 minutes, using an image-based rehabilitation system, by connecting volunteers with a physiotherapist online in their home environment. Telerehabilitation-based motor imagery training will only be applied to the treatment group by the same physiotherapist for 15-20 minutes in addition to the physiotherapy training, three (3) sessions per week for eight (8) weeks.
  Interventions: Procedure: telerehabilitation-based motor imagery training; Procedure: telerehabilitation-based physiotheraphy training
- Group 2 (Active Comparator): Telerehabilitation-based physiotherapy program
  Telerehabilitation-based physiotherapy program; Eight (8) weeks, three (3) sessions per week, 40 minutes, using an image-based rehabilitation system, by connecting volunteers with a physiotherapist online in their home environment.
  Interventions: Procedure: telerehabilitation-based physiotheraphy training
- Healthy children group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Procedure: telerehabilitation-based motor imagery training — Motor imagery is defined as the mental thinking of a movement without actual movement being revealed. Many of the currently available physiotherapy and rehabilitation approaches are designed to stimulate damaged motor neural connections through neuroplasticity.
  based on real movements. Studies have shown that similar brain regions are activated during motor imagery and real movement. By repeatedly visualizing the same movement, people can improve their motor activity skills such as lifting weights, playing the piano or performing surgery. These findings suggest that motor imagery provides motor learning by strengthening synaptic connections depending on activity.
  Arms: Group 1
Procedure: telerehabilitation-based physiotheraphy training — The telerehabilitation application will be carried out by video conference method, one of the image-based telerehabilitation technologies. The telerehabilitation-based physiotherapy program will be administered to both Group 1 and Group 2 children by a physiotherapist experienced in the physiotherapy of neuromuscular diseases, excluding the researchers who performed the randomization and evaluations.
  Arms: Group 1; Group 2

SUMMARY:
When the field of neurorehabilitation is examined, most of the current physiotherapy and rehabilitation approaches are based on real movements to stimulate damaged motor neural connections through neuroplasticity. However, since studies have shown that similar brain regions are activated during real movement with motor imagery, which is defined as imagining movement without actually revealing the movement, the findings of these studies suggest that motor functions can be improved through neuroplasticity, just like real movement. When the literature especially in the pediatric population is examined; The effectiveness of motor imagery training with children with cerebral palsy was examined and positive results were found. However, there are no such studies on children with DMD. In addition, telerehabilitation-based motor imagery training is a very rare treatment modality that requires further research. Therefore, the aim of the study is to investigate the effect of telerehabilitation-based motor imagery training on motor imagery ability, motor function and physical performance in children with DMD. The secondary aim of the study is to investigate the effects of telerehabilitation-based motor imagery training on psychosocial factors including fatigue and quality of life in children with DMD.

DETAILED DESCRIPTION:
The primary aims of this study are;

1. To determine the motor imagery ability in children with DMD and compare it with healthy children,
2. To investigate the effect of telerehabilitation-based motor imagery training on motor imagery ability, motor function and physical performance in children with DMD. The secondary aim of the study is to investigate the effects of telerehabilitation-based motor imagery training on psychosocial factors including fatigue and quality of life in children with DMD.

It is aimed that the data obtained as a result of this study will guide physiotherapists while preparing rehabilitation programs for DMD patients. When the literature is examined, it is reported that motor imagery training is used in many pediatric diseases such as cerebral palsy, brachial plexus, developmental coordination disorder and has positive effects. No study was found in which the effectiveness of motor imagery training was investigated in children with DMD. With this study, it is aimed to contribute to the literature by investigating the effects of motor imagery training to be applied to children with DMD on motor imagery skills, motor function and physical performance.

After determining the functional levels of the children with DMD included in our study according to the Brooke Lower Extremity Functional Classification, a stratified randomization method will be applied by a researcher who was not involved in the evaluation and treatment intervention based on these levels. Thus, patients with DMD will be divided into 2 groups as Group 1 and Group 2. The above-mentioned evaluations of children with DMD will be made twice, before and after the treatment, by a researcher other than the researcher who performed the patient selection and randomization. In order to compare the pre-educational motor imagery skills of children with DMD with healthy children, the group of healthy children will be evaluated only once and no training will be applied to this group.

The interventions to be applied to the groups in the study are summarized below;

Group 1 (children with DMD): Telerehabilitation-based physiotherapy program + telerehabilitation-based motor imagery training

Group 2 (children with DMD): Telerehabilitation-based physiotherapy program

Healthy child group: No intervention will be applied Sessions will be planned three (3) times a week for eight (8) weeks, and session times will be planned by considering the fatigue levels of the children and school hours.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of DMD diagnosis by clinical, diagnostic studies and molecular genetic studies,
* According to Brooke Lower Extremity Functional Classification, it is at Circuit 1-2 levels (early period),
* To be between the ages of 7-15,
* To be able to comply with the physiotherapist's instructions, to have a score of 27 and above (between 27 and 35 indicates normal cognitive level) in the Modified Mini Mental Test,
* Having a computer and an active internet connection at home

Exclusion Criteria:

* Inability to communicate adequately with the physiotherapist,
* In the last 6 months, having deformities that may prevent performance evaluations or physiotherapy program, having any injury and / or surgery of the lower / upper extremities
* Having any additional neurological/orthopedic problems other than DMD

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Duchenne muscular dystrophy (DMD) is an X-linked recessive genetic disorder with a prevalence of approximately 1/3600-6000 live male births.
Enrollment: 36 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Kinesthetic and Visual Imagery Questionnaire (KVIQ)-10 | Change from Baseline at 8 weeks
  Kinesthetic and Visual Imagery Questionnaire-10 is a 10-item version consisting of 5 movements, and each item is scored between 1 and 5 in the same way. The total score of the questionnaire varies between 10-50. The kinesthetic and visual imagery sub-scores range from 5 to 25. High scores indicate good visualization ability.
Movement Imagery Questionnaire for Children (MIQ-C) | Change from Baseline at 8 weeks
  During this test, which is applied with a physiotherapist, children will be asked to physically perform the movement in the items in the instruction once, and then imagine that they are doing the movement from 3 different perspectives. The clarity of these imagery will be scored using a Likert-type scale from 1 (very difficult to feel) to 7 (very easy to feel).
Mental Chronometry Test | Change from Baseline at 8 weeks
  In the mental stopwatch application; Children will be asked to make a movement and then be asked to imagine that movement. In our study, mental chronometer measurements for timed performance tests (standing from supine to standing up, walking 10 meters, climbing 4 steps, descending 4 steps) and the Four Square Step Test (DKAT) will be made with a stopwatch. Simultaneously with the start command, the stopwatch will be started, and the individual will start the imagery of the task and the stopwatch will be stopped as soon as he/she indicates that he/she has finished the imagery.
  The temporal coherence between real and imagined motion will be calculated in terms of delta time with the formula "(real motion-imagined motion)/[(actual motion + imagined motion)/2] x 100".
6 minutes walk test | Change from Baseline at 8 weeks
  participants were instructed to travel as far and as fast as possible in six minutes on 25 meter-indoor course.
Timed performance tests | Change from Baseline at 8 weeks
  Timed function tests included time taken to stand from a supine position, time taken to run 10 m, time taken to climb 4 standard-sized stairs, time taken to descend 4 standard-sized stairs
Four Square Step Test | Change from Baseline at 8 weeks
  Four Square Step Test is performed by asking the child to step clockwise and counterclockwise from square 1 to square 4 against time on a floor that is divided by sticks to form 4 squares and numbered from 1 to 4. It is a timed test measured with a stopwatch. Time starts when the child lifts his or her foot to take a step. Time is stopped when both feet reach square 1 again. The dynamic balance of the child is interpreted by looking at the completion time of the test. Accordingly, shorter test time indicates better dynamic balance.
Motor Function Measurement (MFM) | Change from Baseline at 8 weeks
  The items in this outcome measure, which evaluate functions in 3 different sections (standing and transfers (D1), proximal/axial (D2) and distal (D3)) in a total of 32 items, are scored between 0 and 3. 0; cannot initiate any movement and maintain the starting position, 1; partially completes the move, 2; makes movement slowly and visibly clumsily, with compensations, 3; makes the movement in the specified standard pattern. A score between 0-96 is taken from the scale. High scores indicate higher motor function.
North Star Ambulation Assessment | Change from Baseline at 8 weeks
  Using the NSAA, patients' ambulations are scored with a 3-level grading system as "acting normally without assistance=2", "doing it with compensation=1" and "inability to perform the activity independently=0". It contains 17 items. . The total score ranges between 0-34. A higher score indicates better ambulation and motor function.

SECONDARY OUTCOMES:
PedsQL Multidimensional Fatigue Scale | Change from Baseline at 8 weeks
  The fatigue of children with DMD will be assessed with the PedsQL Multidimensional Fatigue Scale. This scale evaluates fatigue with a total of 18 items, six items under each heading and three main headings as "General Fatigue", "Fatigue in Sleep/Resting" and "Cognitive Fatigue". It has three different forms for young children (5-7 years old), children (8-12 years old) and adolescents (13-17 years old). In the young child report, each item is scored as "Not always=0", "Sometimes=2" and "Very=4", while in other forms, each item is scored 0, 1, 2, with answers ranging from "Never" to "Almost always". It can get 3, 4 points. All three forms have both child and parent reports.
Pediatric Quality of Life Inventory-3.0 (PedsQL-3.0)-Neuromuscular Module | Change from Baseline at 8 weeks
  The Pediatric Quality of Life Inventory-3.0 (PedsQL-3.0)-Neuromuscular Module Turkish version PedsQL-3.0 Neuromuscular Module will be used to evaluate the health-related quality of life of children with DMD. The scale consists of 25 items under 3 categories. Items are scored on a Likert-type scale from 0 (never poses a problem) to 4 (always poses a problem). Scoring is between 0-100 (0 points=100, 1 point=75, 2 points=50, 3 points=25, 4 points=0) at the end of the test. Higher scores on the PedsQL-3.0 Neuromuscular Module indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: İpek Gürbüz, Prof, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Bora-Zereyak M, Bulut N, Yilmaz O, Haliloglu G, Alemdaroglu-Gurbuz I. The effects of telerehabilitation-based motor imagery training on motor imagery ability, motor function and physical performance in Duchenne muscular dystrophy. Disabil Rehabil. 2025 Jul;47(15):3866-3875. doi: 10.1080/09638288.2024.2438251. Epub 2024 Dec 9. PMID 39648851